CLINICAL TRIAL: NCT05869526
Title: A Comparison of the Effects of Krill Oil and Fish Oil Supplementation on Muscle Function in Older Adults: a Randomised Controlled Pilot Study
Brief Title: A Comparison of the Effects of Krill Oil and Fish Oil Supplementation on Muscle Function in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Stuart Gray, Professor, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FISHKRILL
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Sarcopenia
Keywords: muscle mass; strength; omega-3; ageing
MeSH Terms: conditions — Sarcopenia | interventions — Fish Oils; Plant Oils

STUDY DESIGN:
Intervention Model Description: 1:1:1 basis
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Supplements will be identical in look and taste
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fish oil (Active Comparator): Fish oil 4 g/day
  Interventions: Dietary Supplement: Fish oil
- Krill oil (Active Comparator): Krill oil 4g/day
  Interventions: Dietary Supplement: Kril oil
- Placebo (Placebo Comparator): Vegetable oil 4g/day
  Interventions: Dietary Supplement: Vegetable oil

INTERVENTIONS:
Dietary Supplement: Fish oil — EPA rich fish oil
  Arms: Fish oil
Dietary Supplement: Kril oil — Superba Krill Oil
  Arms: Krill oil
Dietary Supplement: Vegetable oil — Mixed vegetable oil
  Arms: Placebo

SUMMARY:
The aim of the study is to compare the effects of Krill Oil and Fish Oil supplementation on muscle function in older adults. The secondary aim is to investigate the mechanisms underlying the beneficial effects previously observed.

ELIGIBILITY:
Inclusion Criteria:

* Older adults (aged 60 years or older). BMI less than 30kg/m2

Exclusion Criteria:

* Participants (diagnosed and being treated for a pre-existing medical condition (cancer, kidney disease, liver disease, diabetes mellitus and cardiovascular disease, uncontrolled hypertension, gait disturbances limiting the ability to perform assessments of muscle function, dementia, affecting muscles known to use drugs (e.g., steroids). History of allergy to fish or fish oil and regular consumption of more than1portion of oily fish per week or use of fish oil or krill oil supplements will also be excluded.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Change in knee extensor maximal isometric torque ( MVC) | Change from baseline to 16 weeks
  Knee extensor maximal isometric torque measured during a maximal voluntary contraction

SECONDARY OUTCOMES:
Change in fat mass | Change from baseline to 16 weeks
  Whole body fat mass measured by measured via bio-electrical impedance
Change in lean mass | Change from baseline to 16 weeks
  Whole body lean mass measured by measured via bio-electrical impedance
Blood sample | Change from baseline to 16 weeks
  Red Blood Cell Omega-3 levels
Change in Grip strength | Change from baseline to 16 weeks
  Grip strength measured with a hand held dynamometer
Change in Muscle thickness | Change from baseline to 16 weeks
  Vastus lateralis muscle thickness measured by ultrasound
Force steadiness during submaximal isometric knee extensor contractions | Change from baseline to 16 weeks
  Measured by using intramuscular iEMG
Neuromuscular Junction (NMJ) | Change from baseline to 16 weeks
  Measured by iEMG
Change in gait speed | Change from baseline to 16 weeks
  Time taken to walk 4 metres at a normal walking pace
Change in Chair rise time | Change from baseline to 16 weeks
  A 30-second sit-to-stand test measured functional abilities

OTHER OUTCOMES:
Step Time (Sec) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Cycle Time (Sec) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Step Length (CM) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Stride Length (CM) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
H-H Base Support (CM) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Single Support (%GC) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Double Support (%GC) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Swing (%GC) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Stance (%GC) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Step/ Extremity Ratio | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Toe In/ Out (deg) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Distance (CM) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Ambulation Time (Sec) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Velocity (CM/Sec) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Mean Normalized Velocity | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Number of Steps | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Cadence (Steps/Min) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Step Time Differential (Sec) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Step Length Differential (CM) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat
Cycle Time Differential (Sec) | Change from baseline to 16 weeks
  Measured during a 4m walk using a gaitrite mat

CONTACTS AND LOCATIONS:
Locations (1):
- Stuart Robert Gray, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No